CLINICAL TRIAL: NCT02572271
Title: Mastopexy With Autologous Augmentation in Women After Massive Weight Loss - A Clinical, Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Peder Ikander, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20150106CKH/bss
Record Dates: First submitted 2015-10-03; First posted 2015-10-08 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Weight Loss
Keywords: Autologous augmentation; Mastopexy; Massive weight loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rubins Mastopexy (Active Comparator): Patients are allocated to a mastopexy using Rubins technique
  Interventions: Procedure: Rubins Mastopexy
- LOPOSAM (Active Comparator): Patients are allocated to a mastopexy using the LOPOSAM technique
  Interventions: Procedure: LOPOSAM

INTERVENTIONS:
Procedure: Rubins Mastopexy — The surgical technique described by Rubin is performed. No other intervention.
  Arms: Rubins Mastopexy
Procedure: LOPOSAM — The surgical technique LOPOSAM is performed. No other intervention.
  Arms: LOPOSAM

SUMMARY:
The purpose of this study is to compare two different techniques of mastopexy with autologous augmentation, the Lower Pole Subglandular Advancement Mastoplasty (LOPOSAM) and Rubins Mastopexy with autologous augmentation, in massive weight loss patients to see if one technique is superior to the other.

DETAILED DESCRIPTION:
In Massive Weight Loss (MWL) patients the breasts often appear deflated following the prominent volume decrease. The breast is not only deflated, the supportive fibrous tissue is lax and the structural properties have changed. In the typical patient the breast base has sunk along with the inframammary crease and the shape of the breast is wide and flat with a significant ptosis.

One way of helping these women is to offer a mastopexy with autologous augmentation. There are several different surgical techniques for treating the ptotic and deflated breast in MWL patients.

In this study the investigators compare the investigators own technique, LOPOSAM, with Rubins Mastopexy with autologous augmentation.

In Rubins Mastopexy, an extensive re-arrangement of the skin, fat and breast tissue is done and this is supposed to give good long term results. The procedure is however time consuming and extensive.

The LOPOSAM technique is less extensive and therefore less time consuming and the investigators hypothesis is therefore that the technique has a lower complication rate.

Women that is referred for mastopexy after MWL and meet the criteria for post bariatric surgery, set by the Danish National Board of Health, and is found to be a suitable candidate for mastopexy with autologous augmentation is invited to participate in the study.

Sample size assessment has shown that 22 women (11 in each group) is needed and this number of patients is expected to be recruited in 6-9 months.

The study design is a prospective randomized trial.

Preoperative breast measurements and clinical photographs will be compared with measurements and clinical photographs at 3, 6 and 12 months postoperative

The primary outcome is operation time but secondary outcomes include economics, breast measurements, cosmetic result and complication rates.

With this trial, the investigators hope to demonstrate whether or not one of the two techniques is superior to the other and therefore should be the preferred technique.

ELIGIBILITY:
Inclusion Criteria:

* Women that meet the Danish National Board of Health criteria for post bariatric surgery, and is found to be a suitable candidate for autologous augmentation

Exclusion Criteria:

* Severe dementia, making informed consent impossible
* Non-Danish speaking

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Operation Time | Intraoperative
  The time of surgery from start to finish is registered for both techniques.

SECONDARY OUTCOMES:
Costs of treatment | 1 year
  In order to evaluate the socio-economic aspects and cost-benefit associated with the use of each surgical technique we record the following parameters for all patients: Duration of operation, duration of hospitalization, duration of entire course of the breast reconstruction, duration of sick leave and need for revisional/correctional procedures. With these data we can evaluate which technique is the most cost beneficial
Breast measurements | 1 year
  Standardized breast measurements preoperative and at 3, 6 and 12 months postoperative is registered. Measurements registered include sternal notch to nipple distance, breast base and height, projection of the breast and ptosis of the breast, measured with a tape measure.
  From this data the investigators can evaluate the long lasting effect of the different techniques
Cosmetic result | 1 year
  The cosmetic result will be evaluated both by the patient on a scale from 1-10 at 3, 6 and 12 months postoperative and by external senior plastic surgeons by evaluating clinical photographs
Complications | 3 months
  Difference in complications between the two techniques will be registered during the follow-up period.They will include: wound dehiscence, partial necrosis, infection and haematoma. Complications will be classified as either major or minor depending on the need for surgical revision

CONTACTS AND LOCATIONS:
Overall Officials: Peder Ikander, MD, Principal Investigator — Department of Plastic and Reconstructive Surgery, Odense University Hospital, Odense, Denmark
Locations (1):
- Odense University Hospital, Department of Plastic and Reconstructive Surgery, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubin JP. Mastopexy after massive weight loss: dermal suspension and total parenchymal reshaping. Aesthet Surg J. 2006 Mar-Apr;26(2):214-22. doi: 10.1016/j.asj.2006.01.010. PMID 19338902
- [Background] Rubin JP, Khachi G. Mastopexy after massive weight loss: dermal suspension and selective auto-augmentation. Clin Plast Surg. 2008 Jan;35(1):123-9. doi: 10.1016/j.cps.2007.08.008. PMID 18061806
- [Background] Gusenoff JA, Rubin JP. Plastic surgery after weight loss: current concepts in massive weight loss surgery. Aesthet Surg J. 2008 Jul-Aug;28(4):452-5. doi: 10.1016/j.asj.2008.06.001. PMID 19083561
- [Background] Rubin JP, Gusenoff JA, Coon D. Dermal suspension and parenchymal reshaping mastopexy after massive weight loss: statistical analysis with concomitant procedures from a prospective registry. Plast Reconstr Surg. 2009 Mar;123(3):782-789. doi: 10.1097/PRS.0b013e31819ba1a8. PMID 19319040
- [Background] Thoma A, Kaur MN, Tsoi B, Ziolkowski N, Duku E, Goldsmith CH. Cost-effectiveness analysis parallel to a randomized controlled trial comparing vertical scar reduction and inverted T-shaped reduction mammaplasty. Plast Reconstr Surg. 2014 Dec;134(6):1093-1107. doi: 10.1097/PRS.0000000000000751. PMID 25255113
- [Background] Hansson E, Manjer J, Ringberg A. Inter-observer reliability of clinical measurement of suprasternal notch-nipple distance and breast ptosis. Indian J Plast Surg. 2014 Jan;47(1):61-4. doi: 10.4103/0970-0358.129625. PMID 24987206
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Fischer JP, Cleveland EC, Shang EK, Nelson JA, Serletti JM. Complications following reduction mammaplasty: a review of 3538 cases from the 2005-2010 NSQIP data sets. Aesthet Surg J. 2014 Jan 1;34(1):66-73. doi: 10.1177/1090820X13515676. Epub 2013 Dec 13. PMID 24334499
- [Background] Cardoso MJ, Cardoso JS, Wild T, Krois W, Fitzal F. Comparing two objective methods for the aesthetic evaluation of breast cancer conservative treatment. Breast Cancer Res Treat. 2009 Jul;116(1):149-52. doi: 10.1007/s10549-008-0173-4. Epub 2008 Sep 7. PMID 18777134
- [Background] Godwin Y, Barron EJ, Edmunds MC, Meyer M, Bardsley A, Logan AM, O'Neill TJ, Wood SH. A comparison of the patient and surgeon opinion on the long-term aesthetic outcome of reduction mammaplasty: have we improved over 15 years? J Plast Reconstr Aesthet Surg. 2014 Jul;67(7):932-8. doi: 10.1016/j.bjps.2014.04.006. Epub 2014 May 9. PMID 24860932
- See also: The Danish National Board of Health criteria for post bariatric surgery — http://sundhedsstyrelsen.dk/da/sundhed/kvalitet-og-retningslinjer/nationale-kliniske-retningslinjer/udgivelser/visitationsretningslinjer/~/media/805344BC849E4050857B85345AC14F39.ashx?m=.pdf